CLINICAL TRIAL: NCT01566370
Title: Zonisamide for Heavy Drinkers With Bipolar Disorder
Acronym: ZNSBP
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: recruitment infeasible
Sponsor: Yale University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZNS-BP; VACT MIRECC (Other: VA); K23AA017689 (NIH)
Record Dates: First submitted 2011-12-15; First posted 2012-03-29 (Estimated); Results first posted 2016-04-22 (Estimated); Last update posted 2017-01-13 (Estimated); Status verified 2016-11

CONDITIONS: Alcohol Use Disorders; Bipolar Disorder
Keywords: alcoholism; alcohol use disorder; alcohol dependence; alcohol abuse; bipolar; anticonvulsant; zonisamide
MeSH Terms: conditions — Alcoholism; Bipolar Disorder | interventions — Zonisamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Zonisamide (Experimental): Subjects will receive zonisamide titrated to a target dose of 500mg orally, daily, double-blind
  Interventions: Drug: Zonisamide
- Placebo (Placebo Comparator): Patients will receive placebo pills that are made to match the zonisamide medication (via over-encapsulation, double-blind, subjects will receive same number of capsules as the active medication group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zonisamide — titration of dose to 500mg oral, daily, over 8 weeks, then 6 weeks of treatment at that dose
  Other Names: Zonegran
  Arms: Zonisamide
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, placebo controlled trial of the medication zonisamide for the purpose of reducing heavy drinking and drinking, as well as reducing mood symptoms, in bipolar subjects that drink excessively and heavily.

Hypotheses: (Primary aims); Add-on zonisamide compared to placebo will result in:

1. significant reduction in heavy drinking days, drinks per week and per drinking day, and significantly greater increase in abstinent days, ii) greater rates of abstinence and abstinence to heavy drinking, greater reduction in biomarkers of heavy alcohol use such as gamma-glutamyl transferase (GGT), and greater reduction in alcohol urge or "craving",
2. Significant reduction in prevalent mood symptoms on the BRMS and BRMeS, CARS, HAMD, or no worsening of euthymic mood, and significant improvement on the Clinical Global Impressions Scale-Severity.
3. (Secondary aims) Add-on zonisamide compared to placebo will result in significant reduction in weight (kilograms) and other secondary weight-related metabolic factors such as fasting glucose, lipid profile, and blood pressure.
4. (Secondary aims) Add-on zonisamide compared to placebo will result in improved clinical global impression, overall functioning, quality of life, and reduced medical symptoms.

5.) (Exploratory Aims) To will examine interactions between genotype and medication on treatment response for allelic variation in genetic loci related to the major neurotransmitter and neurophysiologic pathways that are relevant to bipolar disorder, alcoholism, and zonisamide mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Female/male aged 18-65 years
* Ability to provide informed consent to participate
* Presence of Axis I diagnosis of BD (either type I, Type II, or NOS), in manic, hypomanic, depressive, mixed, or euthymic states plus presence of Axis I diagnosis of a current AUD and/or "at risk" regular heavy drinking (must average >2 heavy drinking days per week) with the goal of reducing or stopping drinking
* treatment with a standard mood stabilizer medication and or other medications with known psychotropic effects on mood state but not alcohol use; Lithium, and/or atypical antipsychotic medications will be the preferred medications,
* Subjects not on any primary acceptable mood stabilizer as described above must be willing to begin treatment with Lithium in open label fashion,
* English speaking, Able to read at the eighth grade or higher level and show no evidence of significant cognitive impairment;
* Women of child-bearing potential (i.e., no hysterectomy, bilateral oophorectomy, or tubal ligation or <2 years postmenopausal), must be non-lactating, practicing a reliable method of birth control, and have a negative serum pregnancy test prior to initiation of treatment;
* Must continue to have at least 2 heavy drinking days per week (averaged per month, with heavy drinking defined as having >4 standard drinks per day for males, and >3 standard drinks per day for females) up to the screening appointment

Exclusion Criteria:

* Presence of another major Axis I disorder such as Schizophrenia or Schizoaffective disorder, Delusional disorder, or other severe psychiatric disorder. A history of suicidal or violent behavior which, in the opinion of the study physician, puts the patient at significant risk of suicide or homicide during the study.
* Past history of drug abuse or dependence will be allowed, but active drug dependence (with the exception of nicotine dependence) in the last 30 days will be disqualifying.
* Serious neurological, or endocrine disorder,
* Evidence of potentially serious or as yet undiagnosed medical problems,
* Neurocognitive cognitive or language limitations, or other incapacity with providing informed consent;
* Known adverse reaction to zonisamide, sulfa-drug allergy, penicillin allergy, other severe adverse drug reaction or allergy, or any serious systemic autoimmune illness,
* Patients currently undergoing ECT treatment.
* Also patients with a history of seizures (other than febrile seizures), renal calculi, or currently taking medications that could either significantly increase the risk of seizures (e.g., tricyclic antidepressant agents, Bupropion, clozaril), or that could potentially theoretically significantly influence drinking behavior such as benzodiazepines, stimulants, opioid painkillers, sedative-hypnotics, etc.).
* Subjects on the following anticonvulsant medications will also be excluded as they may increase the risk of similar side-effects (similar to zonisamide) such as rash, cognitive impairment, or potentially could confound the study of drinking behavior; topiramate, tiagabine, oxcarbazepine, carbamezapine, valproic acid, lamotrigine
* Patients who, on clinical examination by a physician, are deemed to be too severely alcohol dependent to permit them to participate in an outpatient level of care medication trial. We have, over the years, developed methods for reliably and safely assessing patients for alcohol treatment and dual diagnosis studies.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert J Arias, MD, Principal Investigator — Yale University, VA CT Health System
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Zonisamide | Placebo
Started | 2 | 1
Completed | 0 | 0
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Population: Heavy drinkers with bipolar disorder
Groups:
- Total: Total of all reporting groups
Arm/Group | Zonisamide | Placebo | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 58.5 [57 to 60] | 45 [45 to 45] | 51.75 [45 to 60]
Gender [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Total Heavy Drinking Days
Description: The percentage of total heavy drinking days compared between groups (zonisamide and placebo) during the time spent on the target dose of the medication (i.e., not including the titration or taper periods), totaled between the time-points of weeks 11 and 14 (4 weeks time frame).
Time Frame: from week 11 through 14 (over 4 weeks)
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change on Hamilton Depression Rating Scale
Description: Change from baseline to endpoint in Hamilton scores compared between medication and placebo, using repeated measures
Time Frame: 14 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Change in Clinician Assisted Rating Scale for Mania (CARS-M) Scores
Description: Comparison between groups on change in scores on the CARS-M over 14 weeks from baseline to endpoint, measured weekly and analyzed with repeated measures
Time Frame: 14 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Percentage of Abstinent Days
Description: The difference in total percentage of abstinent compared between groups (zonisamide and placebo) during the time spent on the target dose of the medication (i.e., not including the titration or taper periods), which includes week 11, 12, 13, and 14.
Time Frame: over four weeks, from week 11 through 14
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in Alcohol Urge Questionnaire Score
Description: This is the change in AUQ scores (urge to drink) measured weekly compared between groups using repeated measures
Time Frame: from baseline to endpoint, 14 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Gamma Glutamyl Transferase (GGT)
Description: Difference between groups on change in levels of GGT over time, measured at baseline, week 5, week 9, week 13, and endpoint, using repeated measures
Time Frame: 14 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Beck Depression Inventory (BDI) Scores
Description: Comparison between groups on change in BDI scores over the 14 weeks of the study, measured weekly, using repeated measures
Time Frame: 14 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percentage of Total Drinking Days
Description: The percentage of total drinking days compared between groups (zonisamide and placebo) during the time spent on the target dose of the medication (i.e., not including the titration or taper periods), which includes week 11, 12, 13, and 14.
Time Frame: 4 weeks
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change in Number of Heavy Drinking Days Per Week by Time
Description: A comparison between medication and placebo on the measure of number heavy drinking days per week over the course of the study (baseline to endpoint) via interaction with time using repeated measures
Time Frame: 14 weeks (baseline to endpoint)
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Change in Number of Drinks Per Week by Time
Description: Comparison between medication and placebo groups on the change in number of drinks per week via interaction with time (from baseline to endpoint) using repeated measures
Time Frame: 14 weeks (baseline to endpoint)
Population: None of the subjects completed the study or made it to the 12 week endpoint.
Arm/Group | Zonisamide | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: baseline, week 1, week 2
Description: Adverse events reported on the SAFTEE form.
Arm/Group | Zonisamide | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zonisamide (N=2) | Placebo (N=1)
Nervousness (General disorders) | 1 | 1
Feeling Drowsy (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Depressed Mood (Psychiatric disorders) | 2 | 0
Leg Cramps (Musculoskeletal and connective tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0
Decreased Sex Drive (Reproductive system and breast disorders) | 2 | 0
Headache (Nervous system disorders) | 1 | 1
Mood swings (Psychiatric disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Irritability (General disorders) | 2 | 0
Confusion (Psychiatric disorders) | 2 | 0
Memory Problems (Nervous system disorders) | 1 | 0
Difficulty Paying attention (Nervous system disorders) | 1 | 0
Slowed Movements (General disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Swelling feet/ankles (General disorders) | 0 | 1
Gas (Gastrointestinal disorders) | 0 | 1
Gait Disturbance (General disorders) | 0 | 1
Decreased Sweating (Skin and subcutaneous tissue disorders) | 1 | 0
Extreme Thirst (General disorders) | 1 | 0
Loss of Appette (Metabolism and nutrition disorders) | 1 | 0
Rapid Breathing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aggressive Behavior (Psychiatric disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Pain (Reproductive system and breast disorders) | 0 | 1
Chest pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Difficulty Sleeping (Psychiatric disorders) | 1 | 0
Extreme Tiredness (Nervous system disorders) | 1 | 1
Impotence (Reproductive system and breast disorders) | 1 | 0
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No